CLINICAL TRIAL: NCT06100432
Title: Effect of Eurycoma Longifolia (DLBS5055) and Multivitamins (Vitamin C+Vitamin E+ Β-carotene) on Sperm Parameters and Reproductive Hormones of Infertile Males in Yogyakarta, Indonesia
Brief Title: Effect of Eurycoma Longifolia (DLBS5055) and Multivitamins (Vitamin C+Vitamin E+ Β-carotene) for Infertile Males
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duta Wacana Christian University (Other)
Collaborators: Dexa Medica Group (Industry)
Responsible Party: Principal Investigator, dr. Seso Sulijaya Suyono, Sp.And, MD, Duta Wacana Christian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UST00223
Record Dates: First submitted 2023-10-06; First posted 2023-10-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Male Infertility
Keywords: Oligozoospermia
MeSH Terms: conditions — Infertility, Male; Oligospermia | interventions — Geritol; Ascorbic Acid; Vitamin E; beta Carotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment 1 (Experimental): DLBS5055 & Placebo Multivitamin
  Interventions: Drug: DLBS5055 200mg; Drug: Placebo Multivitamin
- Treatment 2 (Active Comparator): Multivitamin (Vitamin C 1000mg + Vitamin E 200IU + Beta Carotene 20000IU) & Placebo DLBS5055
  Interventions: Drug: Placebo DLBS5055; Drug: Multivitamin (Vitamin C 500mg + Vitamin E 100IU + Beta Carotene 10000IU)
- Treatment 3 (Experimental): DLBS5055 & Multivitamin (Vitamin C 1000mg + Vitamin E 200IU + Beta Carotene 20000IU)
  Interventions: Drug: DLBS5055 200mg; Drug: Multivitamin (Vitamin C 500mg + Vitamin E 100IU + Beta Carotene 10000IU)

INTERVENTIONS:
Drug: DLBS5055 200mg — 1x1 caplet
  Other Names: Herbapoten
  Arms: Treatment 1; Treatment 3
Drug: Placebo DLBS5055 — 1x1 caplet
  Other Names: Placebo Herbapoten
  Arms: Treatment 2
Drug: Multivitamin (Vitamin C 500mg + Vitamin E 100IU + Beta Carotene 10000IU) — 1x2 caplets
  Other Names: Oxyvit C+
  Arms: Treatment 2; Treatment 3
Drug: Placebo Multivitamin — 1x2 caplets
  Other Names: Placebo Oxyvit C+
  Arms: Treatment 1

SUMMARY:
Infertility is defined as the inability of a couple to get pregnant after one year of regular and unprotected sexual intercourse. Although it is not a life-threatening condition, infertile couple often suffer from mental health issues, including depression and low self-esteem that may impact their Quality of Life (QoL). Male factors contribute to a half of the underlying causes of infertility and semen analysis play a vital role in investigation of the fertility status of the male partners. By performing semen analysis, we could predict the chance of a couple to conceive.

Male infertility treatments include surgery, hormonal treatment and also assisted reproductive techniques, such as intra uterine insemination and in vitro fertilization that may lead to a financial burden for infertile couple. For facing this issue, traditional or herbal medicine and antioxidants are often be used as an alternative way by many infertile couples. One of the traditional medicines used in Indonesia and other Southeast-Asia Countries for infertility cases is Eurycoma longifolia or Pasak Bumi.

Based on previous studies in animals, Eurycoma longifolia could improve Testosterone and may improve sperm parameters, even though there are very few studies in human including in Indonesia. Antioxidants (multivitamins) are also routinely given to the infertile men as they could protect sperm damages from oxidative stress and may in advanced improve sperm quantity and quality. Our study aims to compare the effect of Eurycoma longifolia, Multivitamins and the combination on sperm parameters and also reproductive hormones of the infertile males.

DETAILED DESCRIPTION:
Study population will be idiopathic infertile males who come to the study site. Those who meet inclusion and exclusion criteria will be randomized into three groups (30 subjects each group). Therefore, it will be total 90 subjects planned to be enrolled in the study.

There will be 3 groups of treatment:

Treatment 1: Eurycoma longifolia (DLBS5055) 200mg caplet Treatment 2: 2 caplets of Multivitamin (each caplet consists of Vitamin C 500mg + Vitamin E 100IU + Beta Carotene 10000IU) Treatment 3: Eurycoma longifolia (DLBS5055) 200mg caplet and 2 caplets of Multivitamin (each caplet consists of Vitamin C 500mg + Vitamin E 100IU + Beta Carotene 10000IU)

Because this study will be double-blind randomized controlled trial, each subject still received 3 caplets (one caplet of DLBS5055 or its placebo and two caplets of multivitamin or their placebo), based on treatment group where the subject will be allocated. DLBS5055 caplet or its placebo will be administered once daily 30 minutes after lunch, whereas two multivitamin caplets will be administered once daily 30 minutes after breakfast.

Eligible subjects will be randomly allocated to receive either Treatment 1, Treatment 2 or Treatment 3 for 12 weeks. Subjects will be instructed to come to the clinic every 6-week interval throughout the 12-week study period (at the end of Week 6 and at the end of Week 12) for treatment evaluation. The semen analysis and reproductive hormonal evaluation will be performed at Baseline and at the End of therapy (Week 12). Additional testosterone level monitoring will be performed in the middle of study period (at the end of Week 6). Adverse events will be monitored at baseline and every follow-up visit including End of study (Week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Male with idiopathic infertility
2. Age 20-45 years
3. Married and try to conceive.
4. Being registered with the Indonesian Social Health Insurance Administration Body (BPJS).
5. Has sperm concentration more than 5 million per mL.
6. Has testosterone level between 350-600 ng/dl.
7. Withdraw from any antioxidant treatment for at least 14 days before the enrollment of the study.
8. Able to understand and provide Informed Consent

Exclusion Criteria:

1. Has a varicocele and other metabolic diseases such as diabetes mellitus.
2. Has a history of surgery or injury in the genital region.
3. Has a history of acute and chronic inflammatory diseases.
4. Has a known allergy to any ingredients of the active or placebo material of the tested drugs (Eurycoma longifolia, Vitamin C, Vitamin E and Beta-carotene).
5. Has a history of hormonal therapy in the last 6 months.
6. Consumes any herbal or traditional medicine.
7. Consumes any medicine contains steroid.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Sperm Concentration measured in million per milliliter of ejaculates by LensHooke X1 PRO at Week 12 | Baseline and Week 12
  LensHooke X1 PRO is a new semen quality analyzer. Its operation based on artificial intelligence optical microscopic (AIOM) technology and has been validated to have a high level of correlation and agreement with manual standard of semen analysis and Computer-Assisted Semen Analyzer (CASA).
  Sperm Concentration, as known as sperm density, is defined as the number of spermatozoa (sperm cell) per milliliter of ejaculates. According to the recent WHO laboratory manual for human semen analysis in 2021, sperm concentration more than 16 million per milliliter of ejaculates is considered normal.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Progressive Sperm Motility measured in percentage (%) by LensHooke X1 PRO at Week 12 | Baseline and Week 12
  LensHooke X1 PRO is a new semen quality analyzer. Its operation based on artificial intelligence optical microscopic (AIOM) technology and has been validated to have a high level of correlation and agreement with manual standard of semen analysis and Computer-Assisted Semen Analyzer (CASA).
  Progressive Sperm Motility refers to the proportion of spermatozoa (sperm cell) that swim progressively in a straight line or in a large circle from the whole sperm cells in ejaculates. It is measured in percentage (%). According to the recent WHO laboratory manual for human semen analysis in 2021, progressive sperm motility more than 30% is considered normal.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Normal Sperm Morphology measured in percentage (%) by LensHooke X1 PRO at Week 12 | Baseline and Week 12
  LensHooke X1 PRO is a new semen quality analyzer. Its operation based on artificial intelligence optical microscopic (AIOM) technology and has been validated to have a high level of correlation and agreement with manual standard of semen analysis and Computer-Assisted Semen Analyzer (CASA).
  Normal Sperm Morphology refers to the proportion of spermatozoa (sperm cell) with the normal form (according to Kruger Strict Morphology Criteria) from the whole sperm cells in ejaculates. It is measured in percentage (%). According to the recent WHO laboratory manual for human semen analysis in 2021, normal sperm morphology more than 4% is considered normal.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Serum Follicle Stimulating Hormone Level was determined using electro-chemiluminescence immunoassay (ECLIA) by COBAS 6000 core and measured in mIU/milliliter | Baseline and Week 12
  Follicle-stimulating hormone (FSH) is a reproductive hormone secreted by the anterior pituitary in response to gonadotropin-releasing hormone (GnRH) from the hypothalamus. It indicates the ability of testis to produce sperm. According to our FSH reagent kit, normal serum FSH level in men is between 1,5-12,4 mIU/milliliter.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Serum Total Testosterone Level was determined using electro-chemiluminescence immunoassay (ECLIA) by COBAS 6000 core and measured in nanogram/deciliter | Baseline, Week 6 and Week 12
  Testosterone is the primary reproductive hormone in male and responsible for producing male sex characteristic, spermatogenesis and fertility. According to our reagent kit, normal serum total testosterone level in men is between 249-836 nanogram/deciliter (ng/dL). Serum total testosterone level will be measured three times (baseline, week 6 and week 12).
  Change 1= (Week 6 Value - Baseline Value) Change 2= (Week 12 Value - Baseline Value)

SECONDARY OUTCOMES:
Spontaneous Pregnancy Rate | Week 12
  Spontaneous or Natural Pregnancy Rate among participants or subjects in each group Spontaneous Pregnancy Rate = number of participants whose partners conceive / total number of participants in the group
Sexual Performance, measured by change from baseline of International Index of Erectile Function-5 (IIEF-5) Score | Baseline, Week 6 and Week 12
  International Index of Erectile Function-5 (IIEF-5) is a widely used diagnostic tool for diagnosing erectile dysfunction (ED). It is a validated self-administered questionnaire with possible score range from 5 to 25, and ED will be classified into five categories based on the scores: severe ED (score 5-7), moderate ED (score 8-11), mild to moderate ED (score 12-16), mild ED (score 17-21) and no ED (score 22-25).
  Change 1= (Week 6 Value - Baseline Value) Change 2= (Week 12 Value - Baseline Value)
Change from Baseline in SGOT (Serum Glutamic Oxaloacetic Transaminase) level was determined using IFCC method by Architect c4000 and measured in Unit per liter (U/L) | Baseline and Week 12
  SGOT (Serum Glutamic Oxaloacetic Transaminase) or Aspartate aminotransferase (AST) is one of the important biomarkers to evaluate liver functions. AST is an enzyme found in muscle, kidney and highest concentration in liver and heart. Elevated levels of AST in human serum indicate hepatocellular damage. Normal AST in male adult is 0-37 U/L.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in SGPT (Serum Glutamic Pyruvic Transaminase) level was determined using IFCC method by Architect c4000 and measured in Unit per liter (U/L) | Baseline and Week 12
  SGPT (Serum Glutamic Pyruvic Transaminase) or Alanine aminotransferase (ALT) is one of the important biomarkers to evaluate liver functions. ALT is an enzyme found mainly in kidney and greater concentration in liver cells. Any injury to liver cells will increase the serum ALT level. Normal ALT in male adult is 0-50 U/L.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Serum Blood Urea Nitrogen/BUN level was determined using urease method by Architect c4000 and measured in mg/dl | Baseline and Week 12
  Blood Urea Nitrogen is a normal waste nitrogen product found in blood that comes from the breakdown of protein from foods. Increase levels of BUN indicates kidney failure. Normal BUN level is 6-20 mg/dl.
  Change = (Week 12 Value - Baseline Value)
Change from Baseline in Serum Creatinine level was determined using enzymatic method by Architect c4000 and measured in mg/dl. | Baseline and Week 12
  Creatinine is the major metabolic product of protein. It is formed in muscles and excreted through kidney. Increase levels of creatinine indicates problems in kidney function due to several condition. Normal serum creatinine level is 0.67-1.17 mg/dl.
  Change = (Week 12 Value - Baseline Value)

CONTACTS AND LOCATIONS:
Overall Officials: Seso S Suyono, MD, Principal Investigator — Duta Wacana Christian University
Locations (1):
- Laboratorium Klinik Pramita, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zohman GL, Watts HG. Is a routine radiological consultation cost-effective for pediatric orthopedic radiographs? J Pediatr Orthop. 1998 Jul-Aug;18(4):549-51. PMID 9661871
- [Background] Moskovko VM. [Circadian rhythm of blood clotting processes]. Voen Med Zh. 1986 May;(5):57. No abstract available. Russian. PMID 3739276
- [Background] Zuckerman M. P-impulsive sensation seeking and its behavioral, psychophysiological and biochemical correlates. Neuropsychobiology. 1993;28(1-2):30-6. doi: 10.1159/000118996. PMID 8255407
- [Background] Senciall IR, Rahal S, Sethumadhavan K. Solubilisation and fractional precipitation of a steroid alpha-ketol oxidase. J Steroid Biochem. 1985 Dec;23(6A):1083-5. doi: 10.1016/0022-4731(85)90072-x. PMID 4094415